CLINICAL TRIAL: NCT01365143
Title: Prospective Randomized Trial Comparing Robotic Versus Open Radical Prostatectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closing due to slow enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: R. Houston Thompson, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002288
Record Dates: First submitted 2011-05-26; First posted 2011-06-03 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Prostatic Neoplasms; Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

ARMS (2):
- Open Radical Prostatectomy (Active Comparator)
  Interventions: Procedure: Open Radical Prostatectomy
- Robotic radical prostatectomy (Active Comparator)
  Interventions: Procedure: Robotic Radical Prostatectomy

INTERVENTIONS:
Procedure: Robotic Radical Prostatectomy — Robotic assisted radical prostatectomy
  Arms: Robotic radical prostatectomy
Procedure: Open Radical Prostatectomy — Open radical prostatectomy
  Arms: Open Radical Prostatectomy

SUMMARY:
To date, no study has prospectively compared open versus robotic radical prostatectomy in a randomized fashion for patients with prostate cancer. For patients with newly diagnosed prostate cancer who choose surgical management, the choice of surgical approach is often limited to surgeon preference and experience. This study will prospectively randomize patients with localized prostate cancer who are candidates for surgical management to open versus robotic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the prostate
* Deemed a surgical candidate for a bilateral nerve bundle preservation
* Potent
* Continent of urine
* Surgical candidate for both open and robotic nerve-sparing radical prostatectomy
* Age >18

Exclusion Criteria:

* Previous treatment of prostate cancer (radiation, hormones, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Trifecta | at 2 years
  Free from biochemical recurrence, continent, and potent 2 years after radical prostatectomy

SECONDARY OUTCOMES:
Continence | at 3, 12, and 24 months
  Continent of urine
Potency | at 3, 12, and 24 months
  Satisfactory erections
Free from biochemical recurrence | at 3, 12, and 24 months
  PSA <0.2 ng/mL
Acute complications | Within 30 days of surgery
  Any complication according to Calvien classification
Long-term complication | >30 days
  bladder neck contracture, lymphocele
Estimated blood loss | Participants will be followed for the duration of the operation, an expected average of 3 hours
Operative time | Participants will be followed for the duration of the operation, an expected average of 3 hours
Length of hospital stay | Participants will be followed for the duration of the hospital stay, an expected average of 1-2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States